CLINICAL TRIAL: NCT04608708
Title: A Retrospective Radiological Analysis of Cemento-Osseous Dysplasia Using 3D Imaging
Brief Title: 3D Analysis of Cemento-Osseous Lesions
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, assistant professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2020/189
Record Dates: First submitted 2020-10-21; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Bone Diseases; Cone-beam Computed Tomography; Florid Cemento-osseous Dysplasia
Keywords: Bone Diseases; Cone-beam computed tomography; Florid cemento-osseous dysplasia
MeSH Terms: conditions — Bone Diseases; Florid cemento-osseous dysplasia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1. Periapical Cemento-Osseous Dysplasia: In Periapical Cemento-Osseous Dysplasia , the lower anterior teeth are usually affected. In these lesions, normal bone is replaced by fibrous tissue that contains amorphous vascularised calcifications. In the early stage, it can mimic a periapical lesion, but it is usually associated with vital teeth, without any clinical complaint, and it requires no intervention. Histopathologically, the lesion is similar to fibrous dysplasia and ossifying fibroma.
  Interventions: Other: The data of patients who had applied to the clinic for various reasons and were diagnosed with fibro-osseous lesions
- Group 2. Focal Cemento-Osseous Dysplasia: It occurs in a single area of the posterior teeth. Its radiographic and histolopathological features are similar to Periapical Cemento-Osseous Dysplasia
  Interventions: Other: The data of patients who had applied to the clinic for various reasons and were diagnosed with fibro-osseous lesions
- Grup 3. Florid Cemento-Osseous Dysplasia: When the lesions involve two or more quadrants of the jaw, it is defined as Florid Cemento-Osseous Dysplasia. Its radiographic and histolopathological features are similar to Periapical Cemento-Osseous Dysplasia
  Interventions: Other: The data of patients who had applied to the clinic for various reasons and were diagnosed with fibro-osseous lesions

INTERVENTIONS:
Other: The data of patients who had applied to the clinic for various reasons and were diagnosed with fibro-osseous lesions — lesions diagnosed radiologically and followed up for at least one year were included in this study with the help of cone beam computed tomography.

SUMMARY:
COD lesions effect a wide range of different anatomical areas, show different volume and morphometric characteristics.

DETAILED DESCRIPTION:
Fibro-osseous lesions of the jaws are one of the important lesion groups for which identification and diagnosis create clinical difficulties. In previous studies, the features of the lesions and the effects of COD on anatomical structures were analysed via CBCT images by measuring the lesion's dimensions linearly for the first time in the Brazilian population. However, 3D measurements of the volume need to be taken to assess the actual spread over adjacent anatomical structures. The purpose of this retrospective study is to measure the volume of the lesions that have been diagnosed as COD in the Turkish population by using 3D images. This will contribute to an advanced study conducted on the global population to observe a change in these morphologies with respect to different geographical and ethnic origins.

ELIGIBILITY:
Inclusion Criteria:

* They were diagnosed with fibro-osseous lesions with the help of cone beam computed tomography between 2017 and 2020 were included in the study.
* The lesions diagnosed radiologically and followed up for at least one year were included in this study.

Exclusion Criteria:

-Radiographs with insufficient diagnostic images were not included.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: diagnosed with fibro-osseous lesions with the help of cone beam computed tomography between 2017 and 2020 were included in the study
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
the correlation between presence of cemento osseous dysplasia and gender/ age | for three months from the beginning of the study
  It usually affects female and black patients. Most of the patients are initially diagnosed between the ages of 30 and 50, and the diagnosis is almost never made in individuals younger than 20
cemento osseous dysplasia lesion's location and relationship with the anatomical structures | for three months from the beginning of the study
  If the lesions were in association with the teeth, the teeth numbers were recorded. The periphery of the lesions was divided into two sections: well-defined (corticated, sclerotic, non-corticated and partially corticated) and ill-defined (perforating, diffuse and invasive). The shape of the lesion was classified as circular, oval or irregular. The presence of a hypodense capsule was assessed as present, absent or partially present. The involvement with the adjacent structures - cortical bone (lingual and buccal), mandibular canal, mental foramen, nasopalatinal canal, incisive foramen, maxillary sinus, nasal fossa and anterior mandibular canal - was assessed and recorded. The effects on the cortical bone were assessed as intact, thinning, expansion and thinning, thinning and perforation, expansion, thinning and perforation or perforation. The internal calcified parts of the lesions.
cemento osseous dysplasia lesions dimensional measurement of the lesions | for three months from the beginning of the study
  The internal calcified parts of the lesions and the total volume of the lesions were also assessed.
  The greatest linear dimension of the buccolingual, buccopalatinal and mesiodistal positions was measured on the axial plane, while the supero-inferior dimension was measured on sagittal or cross-sectional images.
cemento osseous dysplasia lesions volume of the lesions | for three months from the beginning of the study
  The internal calcified parts of the lesions and the total volume of the lesions were also assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Nil Günaçar, Principal Investigator — Recep Tayyip Erdogan University Training and Research Hospital
Locations (1):
- Recep Tayyip Erdogan University Training and Research Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
e-identified individual participant data for all measures will be made available
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available 5 years after publication
Access Criteria: Data access requests will be reviewed by authors.

REFERENCES:
- [Background] Kato CNAO, Barra SG, Amaral TMP, Silva TA, Abreu LG, Brasileiro CB, Mesquita RA. Cone-beam computed tomography analysis of cemento-osseous dysplasia-induced changes in adjacent structures in a Brazilian population. Clin Oral Investig. 2020 Aug;24(8):2899-2908. doi: 10.1007/s00784-019-03154-x. Epub 2020 Feb 19. PMID 32076867
- [Background] Kato CN, Barra SG, Pereira MJ, Gomes LT, Amaral TM, Abreu LG, Brasileiro CB, Mesquita RA. Mandibular radiomorphometric parameters of women with cemento-osseous dysplasia. Dentomaxillofac Radiol. 2020 May 1;49(4):20190359. doi: 10.1259/dmfr.20190359. Epub 2019 Dec 20. PMID 31846355